CLINICAL TRIAL: NCT03398109
Title: Customized Toric Intraocular Lens Implantation in Eyes With Cataract and Corneal Astigmatism After Deep Anterior Lamellar Keratoplasty (DALK): a Prospective Study
Brief Title: Effectiveness of Toric Intraocular Lenses for Treating Corneal Astigmatism in Patients With Cataract and Previous DALK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Responsible Party: Principal Investigator, Mario Stirpe, Director Clinical Research, Fondazione G.B. Bietti, IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N. 24/15/FB
Record Dates: First submitted 2018-01-07; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Corneal Astigmatism in Cataract Patients and Previous DALK

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Customized toric IOL (Experimental): Customized toric IOL for post-Dalk atigmatism in cataract patients
  Interventions: Device: Customized toric IOL for post-DALK atigmatism

INTERVENTIONS:
Device: Customized toric IOL for post-DALK atigmatism

SUMMARY:
the purpose of this study was to assess the efficacy of custom made toric intraocular lens implantation in patients with simultaneous post-DALK high corneal astigmatism and cataract.

DETAILED DESCRIPTION:
Patients undergoing cataract surgery after DALK for keratoconus were enrolled. Total corneal astigmatism (TCA)was assessed by a rotating Scheimpflug camera combined with Placido disk corneal topography (Sirius; CSO, Firenze, Italy). A customized toric IOL (FIL 611 T, Soleko) was implanted in all eyes. One year postoperatively, refraction was measured, the IOL position was recorded, and vectorial and non-vectorial analysis were performed to evaluate the correction of astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Corneal suture removal had been performed in all cases at least 1 year before cataract surgery.

Corneal astigmatism was stable at least since 6 months before the cataract surgery

Exclusion Criteria:

* other ocular pathologies as glaucoma, retinal disease.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Measure postoperative refractive astigmatism | 6 months
  Postoperative refractive astigmatism expressed in diopters and measured with refraction examination

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Schiano-Lomoriello, MD, Study Director — Fondazione G.B. Bietti

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schiano Lomoriello D, Savini G, Naeser K, Colabelli-Gisoldi RM, Bono V, Pocobelli A. Customized Toric Intraocular Lens Implantation in Eyes with Cataract and Corneal Astigmatism after Deep Anterior Lamellar Keratoplasty: A Prospective Study. J Ophthalmol. 2018 Jul 3;2018:1649576. doi: 10.1155/2018/1649576. eCollection 2018. PMID 30057802